CLINICAL TRIAL: NCT07000305
Title: Cetuximabβ Combined With Envolimab and mFOLFOX6 as First-line Treatment for RAS/BRAF Wild-type, MSS, Unresectable , Metastatic Colorectal Cancer: A Single-arm, Multi-center, Phase II Trail
Brief Title: A Study of Cetuximabβ Combined With Envolimab and mFOLFOX6 in Subjects With Advanced Colorectal Cancer
Acronym: SUPβORT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tao Zhang (Other)
Responsible Party: Sponsor-Investigator, Tao Zhang, Director, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Organization: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMA-CRC-004
Record Dates: First submitted 2025-05-29; First posted 2025-06-02 (Actual); Last update posted 2025-06-02 (Actual); Status verified 2025-05

CONDITIONS: Advanced Colorectal Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- experimental group (Experimental): All subjects meeting the enrollment criteria will receive 8-12 cycles of induction phase treatment with envolimab in combination with cetuximab beta and mFOLFOX6 regimen, and enter into maintenance therapy after assessment of no disease progression, with maintenance regimen of envolimab in combination with cetuximabβ and a fluorouracil-based chemotherapeutic agent (selected by the investigator)
  Interventions: Drug: Cetuximabβ combined with Envolimab and mFOLFOX6

INTERVENTIONS:
Drug: Cetuximabβ combined with Envolimab and mFOLFOX6 — Envolimab, 200 mg, sc, day 1; Cetuximabβ 500 mg/m2 IV over 60- 120 min, day 1; chemotherapy mFOLFOX6; with the above regimen every 14 days for 1 treatment cycle. Then patients who did not experience disease progression within 8-12 cycles were entered into maintenance therapy, which consisted of a fluorouracil-based-chemotherapy with Cetuximabβ and Envolimab regimen until progression or unacceptable toxicity.

SUMMARY:
A study of Cetuximabβ combined with Envolimab and mFOLFOX6 in Subjects with Advanced Colorectal Cancer

ELIGIBILITY:
Inclusion Criteria:

1. have agreed and signed an informed consent form (ICF) and are willing and able to comply with planned visits, study treatments, laboratory tests and other experimental procedures.
2. At the time of signing the ICF, patients must be ≥18 years of age and have a life expectancy of ≥12 weeks in either males or females.
3. Histologically or cytologically confirmed RAS and BRAF wild-type, MSS type colorectal adenocarcinoma.
4. Advanced or metastatic colorectal cancer (AJCC/UICC stage IV) clearly defined by imaging, with at least one measurable lesion that meets the requirements of the criteria for evaluating the efficacy of solid tumors (RECIST version 1.1).
5. no prior systemic therapy (including epidermal growth factor receptor inhibitors such as cetuximab or panitumumab, vascular endothelial growth factor inhibitors such as bevacizumab, immune checkpoint inhibition such as anti-PD-1 or PD-L1 antibodies, and anti-CTLA-4 antibodies) directed against advanced or metastatic colorectal cancer, but are allowed to receive a maximum of one cycle of the mFOLFOX6 regimen prior to enrollment ; Adjuvant/neoadjuvant therapy is considered a first-line systemic therapy for advanced or metastatic disease if recurrence or metastasis occurs during or within 6 months of completion of adjuvant or neoadjuvant chemotherapy.
6. an Eastern Cooperative Oncology Group (ECOG) physical status score of 0-1.
7. have appropriate organ function during the screening period:
8. Female subjects of childbearing potential must have a negative serum pregnancy test within 3 days prior to initiation of study drug administration and be willing to use a medically approved highly effective contraceptive measure (e.g., IUD, birth control pills, or condoms) during the study period and for 3 months after final study drug administration; for male subjects whose partner is a female of childbearing potential, he/she should be surgically sterilized or agree to use a medically approved highly effective contraceptive measure (e.g., IUD, birth control pills, or condoms) during the study period and for 3 months after final study drug administration. 3 months after the final study dose.
9. Participation in other clinical trials during the study period is not permitted.

Exclusion Criteria:

1. previous or concurrent other active malignancies (except for malignancies that have been curatively treated and have been free of morbidity for more than 5 years or carcinoma in situ that can be cured by adequate treatment).
2. Current gastrointestinal diseases such as duodenal ulcer, ulcerative colitis, intestinal obstruction, or other conditions that may cause gastrointestinal bleeding or perforation as determined by the investigator.
3. Thrombotic or embolic events such as cerebrovascular accidents (including transient ischemic attacks), pulmonary embolism, deep vein thrombosis within 12 months prior to enrollment in the study.
4. Myocardial infarction, severe/unstable angina pectoris, NYHA class 2 or higher cardiac insufficiency, clinically significant supraventricular or ventricular arrhythmia, and symptomatic congestive heart failure within 12 months prior to study entry.
5. systemic antibiotic use for ≥ 7 days within 4 weeks prior to study entry or unexplained fever > 38.5°C during screening/prior to first dose (fever due to oncologic causes is eligible for enrollment at the discretion of the investigator).
6. Presence of hydrothorax, ascites, or pericardial effusion uncontrolled with effective therapy within 14 days prior to study entry.
7. Presence of any prior treatment-induced, unabated adverse event Common Terminology Criteria for Adverse Events (NCI CTCAE version 5.0) Grade 2 or greater toxicity (excluding anemia, alopecia, and skin hyperpigmentation).
8. Presence of interstitial lung disease, non-infectious pneumonia, or uncontrolled systemic disease (e.g., diabetes mellitus, hypertension, pulmonary fibrosis, and acute pneumonia).
9. Human Immunodeficiency Virus (HIV) infection or known Acquired Immune Deficiency Syndrome (AIDS), untreated active hepatitis (Hepatitis B, defined as HBV-DNA ≥ 500 IU/ml; and Hepatitis C, defined as HCV-RNA above the lower limit of detection of the analytical method) or co-infection with Hepatitis B and Hepatitis C.
10. Known or suspected history of allergy to any of the drugs of interest used in the study.
11. Pregnant or lactating women.
12. Women of childbearing potential (< 2 years after last menstrual period) or men of childbearing potential who are not using or refuse to use an effective non-hormonal contraceptive.
13. Presence of other serious physical or mental illnesses or abnormal laboratory tests that may increase the risk of participation in the study or interfere with the study results, as well as patients who, in the opinion of the investigator, are not suitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2027-05-20 (Estimated); Study Completion 2028-05-20 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Through out the study (up to 2 years)
  The efficacy of solid tumors was evaluated according to RECIST v1.1

SECONDARY OUTCOMES:
Objective response rate (ORR) | Through out the study (up to 2 years)
  The efficacy of solid tumors was evaluated according to Response Evaluation Criteria in Solid Tumours Version 1.1 (RECIST v1.1).
disease control rate (DCR) | Through out the study (up to 2 years)
  The efficacy of solid tumors was evaluated according to RECIST v1.1
No Evidence of Disease, NED | Through out the study (up to 2 years)
  Percentage of all subjects who received study treatment with no evidence of tumor presence by current investigations (pathology, imaging, molecular biology, etc.).
Overall survival (OS) | Through out the study (up to 2 years)
  The efficacy of solid tumors was evaluated according to RECIST v1.1
Adverse Event (AE), Treatment-Emergent AE (TEAE), Adverse Event of Special Interest (AESI) and Serious Adverse Event (SAE) | Through out the study (up to 2 years)
  Adverse events will be assessed by investigator(s) according to Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE v5.0).

OTHER OUTCOMES:
Predictive biomarkers of clinical response | Through out the study (up to 2 years)
  An assay based on the Olink platform Target 96 Inflammation Panel was performed to analyze protein markers associated with efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University Hospita, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No